CLINICAL TRIAL: NCT00631124
Title: A Double-blind, Randomized, Uncontrolled Study to Evaluate Inhibition of Ovulation of Two Oral Estradiol / Drospirenone Regimens in Healthy Young Female Volunteers Over a Period of 3 Treatment Cycles
Brief Title: A Study to Evaluate Inhibition of Ovulation of Two Oral Estrogen/Progestogen Regimens in Healthy, Young Females Over a Period of 3 Treatment Cycles
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 91697; 2007-004544-73 (EudraCT Number); 311623 (Other: Company internal)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Contraception
Keywords: Contraception
MeSH Terms: interventions — Estradiol; drospirenone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: BAY86-4891 (Estradiol / Drospirenone)
- Arm 2 (Experimental)
  Interventions: Drug: BAY86-4891 (Estradiol / Drospirenone)

INTERVENTIONS:
Drug: BAY86-4891 (Estradiol / Drospirenone) — Monophasic regimen containing estrogen and progestin 1 pre-treatment cycle, 3 treatment cycles
  Arms: Arm 1
Drug: BAY86-4891 (Estradiol / Drospirenone) — Triphasic regimen containing estrogen and progestin 1 pre-treatment cycle, 3 treatment cycles
  Arms: Arm 2

SUMMARY:
Investigation of a new pill containing an estrogen and a progestin in order to monitor the inhibition of the ovulation in young healthy females over 3 treatment cycles

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers,
* Age 18 - 35 years

Exclusion Criteria:

* Contraindications for use of a combined (estrogen/progestogen) contraceptive (e.g. history of venous/arterial thromboembolic disease)
* Regular intake of medication
* Clinically relevant findings (ECG, blood pressure, physical, gynecological examination, laboratory examination)
* Anovulatory pre-treatment cycle

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable will be the proportion of volunteers with ovulation in at least one of the treatment cycles 2 and 3, based on the binary variable ovulation (i.e. Hoogland score 6) with the levels yes and no | 12 months

SECONDARY OUTCOMES:
Assessment of ovarian activity in treatment cycles 2 and 3 | 12 months
Course of gonadotropins (FSH, LH) | 12 months
Endometrial growth | 12 months
Pharmacokinetics of estrogen and progestin in treatment cycle 3 | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/